CLINICAL TRIAL: NCT00284570
Title: ProCalcitonin in the Pediatric Surgical Patient, Evaluation of a New Marker of Infection
Brief Title: Pro-Calcitonin Levels Following Pediatric Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Kevin O. Maher, MD, Associate Prefessor of Pediatrics, Emory University
Other Study IDs: IRB00002022
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Congenital Heart Disease; Sepsis; Infection
Keywords: pediatrics; congenital heart disease; cardiac; cardiopulmonary bypass; infection; sepsis; postoperative; marker for infection; inflammation; cardiac surgery
MeSH Terms: conditions — Heart Defects, Congenital; Sepsis; Infections; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are collected in order to get the procalcitonin level.
Oversight: Data Monitoring Committee: No

SUMMARY:
First, we, the researchers, hope to find out the PCT response to heart surgery in children by taking blood before surgery and each day for four days after surgery. These blood draws will help us figure out the typical Procalcitonin (PCT) response, the normal increase in PCT after heart surgery, and when the PCT level returns to baseline.

Second, we, the researchers, hope to determine the accuracy of PCT as a marker of infection.

Hypothesis

Our hypothesis is that Procalcitonin is superior to other currently used markers of infection and will prove to be a clinically useful tool for evaluation of infection in children following cardiac surgery.

DETAILED DESCRIPTION:
In this research study, we want to look at the difficulty in identifying infections in children who have heart surgery. We also want to look at differentiating between actual infections and the normal post-surgery course that patients go through. We use a number of tools in the Intensive Care Unit to pick out children at risk for an infection. These tools are the physical examination, a fever, white blood cell count, and C-reactive Protein (CRP) level. When a patient has an infection, they usually have a fever, have a high white blood cell count, and have an increased CRP level. However, these are not always correct. The identification of infection remains a challenge and the laboratory markers of infection (white blood cell count and CRP) that are used now are not perfect.

A new marker of infection, Procalcitonin (PCT), has been found and has been tested in adults and children. PCT has recently been approved by the Food and Drug Administration (FDA) as a marker of infection. PCT has been shown to be a more accurate marker of infection for some groups of patients.

Prior work on a small number of children shows that PCT increases shortly just from heart surgery itself, even without infection. There is little information published about how accurate PCT is for identifying infection in the child heart population. In order to use PCT in our patients, we need to know what the normal levels of PCT are after surgery. Thus, when an infection does happen, we can identify it. We also need to take PCT levels when patients are thought to have infections. We will then need to watch for an infection over the next few days to see if the PCT level rises and can actually predict the presence an infection.

Goals:

1. Determine the Procalcitonin response to cardiopulmonary bypass in children undergoing open-heart surgery. Cardiopulmonary bypass causes a pro-inflammatory state in the patient, and associated rise in Procalcitonin. The ability to use PCT as a marker for infection will require knowledge of its typical response to bypass and the time course to return to baseline.
2. Determine the accuracy of Procalcitonin as a marker of infection, and to compare and contrast these findings with currently used laboratory markers.

Specific Aims

1. Evaluate PCT in the postoperative pediatric cardiac surgical patient as a marker for infection and sepsis.
2. Evaluate PCT's response to cardiopulmonary bypass, and as a predictor of outcome following cardiac surgery.
3. Compare PCT to other markers of inflammation and infection (C-reactive protein and white blood cell response).

By doing this study, we hope to find out two things. First, we hope to find out the PCT response to heart surgery in children by taking blood before surgery and each day for four days after surgery. These blood draws will help us figure out the typical PCT response, the normal increase in PCT after heart surgery, and when the PCT level returns to baseline.

Second, we hope to determine the accuracy of PCT as a marker of infection. Whenever we think a patient may have an infection, it is routine care to take some blood and run lab tests such as a white blood cell count, blood culture, and a C-reactive protein level. Patients in the study will also have an additional 10 drops of blood taken for a PCT level at the same time as the routine blood draw. Even though patients may show signs of an infection, the routine blood test do not always come back positive for an infection. We will compare the routine blood test results (positive or negative for an infection) with the PCT level taken at the same time. If most patients with an infection also have a rise in PCT and those patients without an infection have a normal PCT, then we will prove that PCT is a good, accurate marker for infection in our patients.

This research will help us study infection in our patients. It will help distinguish patients with infection, what the risk factors are, how they are treated, and the response to infection. This information will potentially allow us to use an improved test for identifying infection in a high-risk population of children. Patients in the research project will continue to receive the standard of care treatment after heart surgery and there will be no changes in their care during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital heart disease
* Undergoing cardiopulmonary bypass and cardiac surgery
* Newborn (full term) to up to 6 years of age

Exclusion Criteria:

* Premature (less than 37 weeks)
* 6 years of age or older
* Intercurrent illness at time of surgery
* Orthotopic organ transplant recipient
* Pre-operative extra-corporeal support (ECMO)
* Acquired heart disease

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study patients will be recruited from Children's Healthcare of Atlanta at Egleston. The patients will be in the pre-operative clinic, Cardiac Intensive Care Unit or the Cardiac Stepdown Unit.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2006-01; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maher, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] Martin GS, Mannino DM, Eaton S, Moss M. The epidemiology of sepsis in the United States from 1979 through 2000. N Engl J Med. 2003 Apr 17;348(16):1546-54. doi: 10.1056/NEJMoa022139. PMID 12700374
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Background] Hauser GJ, Chan MM, Casey WF, Midgley FM, Holbrook PR. Immune dysfunction in children after corrective surgery for congenital heart disease. Crit Care Med. 1991 Jul;19(7):874-81. doi: 10.1097/00003246-199107000-00009. PMID 2055075
- [Background] Jarvis WR, Edwards JR, Culver DH, Hughes JM, Horan T, Emori TG, Banerjee S, Tolson J, Henderson T, Gaynes RP, et al. Nosocomial infection rates in adult and pediatric intensive care units in the United States. National Nosocomial Infections Surveillance System. Am J Med. 1991 Sep 16;91(3B):185S-191S. doi: 10.1016/0002-9343(91)90367-7. PMID 1928163
- [Background] Mayhall CG. Diagnosis and management of infections of implantable devices used for prolonged venous access. Curr Clin Top Infect Dis. 1992;12:83-110. No abstract available. PMID 1642805
- [Background] Galetto-Lacour A, Zamora SA, Gervaix A. Bedside procalcitonin and C-reactive protein tests in children with fever without localizing signs of infection seen in a referral center. Pediatrics. 2003 Nov;112(5):1054-60. doi: 10.1542/peds.112.5.1054. PMID 14595045